CLINICAL TRIAL: NCT01402596
Title: Evaluation of Pediatric Procedural Sedation With Rectal Chloral Hydrate or Intranasal Midazolam - a Randomized Controlled Trial
Brief Title: Evaluation of Pediatric Procedural Sedation With Rectal Chloral Hydrate or Intranasal Midazolam
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Institution decided on starting a new protocol of sedation, with another methods and that´s why this study has not started.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Eduardo Mekitarian Filho, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: USP-Sed-001
Record Dates: First submitted 2011-07-19; First posted 2011-07-26 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2011-07

CONDITIONS: Traumatic Brain Injury; Computed Tomography; Procedural Sedation
Keywords: Deep Sedation; Pediatrics; Emergency Hospital Services; Midazolam; Chloral hydrate; Randomized controlled trial
MeSH Terms: conditions — Brain Injuries, Traumatic; Emergencies | interventions — Midazolam; Chloral Hydrate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloral hydrate (Active Comparator): Children undergoing CT scanning will receive in this arm 50 mg per kg of rectal chloral hydrate.
  Interventions: Drug: Chloral Hydrate
- Midazolam (Active Comparator): Children undergoing CT scanning will receive in this arm 0,4 mg/kg of nasal midazolam.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — 0,4 mg per kg - intranasal midazolam - once
  Arms: Midazolam
Drug: Chloral Hydrate — 50 mg per kg, rectal
  Arms: Chloral hydrate

SUMMARY:
Thousands of children receive sedation for diagnostic and therapeutic interventions annually, and this number is expected to increase. Children are at higher risk for sedation-related complications than adults. In different scenarios, multiple drugs are used to achieve sedation, each one with particular adverse events that must be monitored and reported.

Children that need CT scans for traumatic brain injuries often need sedation, without needing and IV line for that. Chloral hydrate is an hypnotic agent used since 1832 with low incidence of adverse events; however, despite its worldwide use, it's being abandoned due to bitter taste, long time of sedation onset, vomiting and mild sedation. Intranasal midazolam, on the other hand, produces high and fast concentrations on CSF with greater rates of success but probably with higher adverse events. There are no prospective studies with large series of patients using intranasal midazolam.

The aim of this study is to determine if nasal midazolam is a safer approach and more effective sedative regimen when compared to rectal chloral hydrate to children undergoing CT scans.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing CT scanning for TBI

Exclusion Criteria:

* epistaxis
* suspected or confirmed skull or nasal fracture
* Moderate to severe traumatic brain injury
* hemodynamically unstable

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Participants will be followed for the duration of hospital (emergency department) stay, an expected average of 2-3 hours
  Such as hypoxemia, respiratory depression, vomiting, hypotension

SECONDARY OUTCOMES:
Efficacy of both drugs | Participants will be followed for the duration of hospital (emergency department) stay, an expected average of 2-3 hours
  Patients vital signs and adverse events will be monitored through patient stay in the emergency department. Mean time after sedation is about three hours.
  Variables collected include Ramsay score for sedation. To consider hospital discharge, we will try to validate Aldrette score and compare the scores between the two arms. Mean time to onset of sedation and time of emergency department stay will also be compared as a mark of efficacy of these two drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Mekitarian Filho, MSc, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil